CLINICAL TRIAL: NCT02910167
Title: Observational Prospective Cohort Study to Evaluate the Incidence of Adverse Events (AE), Risk Factors, and Drug Utilization Patterns Related to Treatment With BUSCAPINA COMPOSITUM N From March to December 2016 in Patients From Metropolitan Lima
Brief Title: Observational Prospective Study to Evaluate AEs, Risk Factors and Drug Utilization of BUSCAPINA COMPOSITUM N in Adults From Metropolitan Lima
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 218.705
Record Dates: First submitted 2016-08-30; First posted 2016-09-21 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Acute Pain; Dysmenorrhea
MeSH Terms: conditions — Acute Pain; Dysmenorrhea | interventions — Butylscopolammonium Bromide; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Men with spasmodic syndromes: Men with any type of gastrointestinal, hepato-biliary, urinary or genital spasmodic syndromes
  Interventions: Drug: Hyoscine n-butylbromide; Drug: Paracetamol
- Women with spasmodic syndromes: Women with any type of gastrointestinal, hepato-biliary, urinary or genital spasmodic syndromes
  Interventions: Drug: Hyoscine n-butylbromide; Drug: Paracetamol

INTERVENTIONS:
Drug: Hyoscine n-butylbromide — Hyoscine n-butylbromide 10 mg
  Groups: Men with spasmodic syndromes
Drug: Paracetamol — Paracetamol 500 mg
  Groups: Men with spasmodic syndromes
Drug: Hyoscine n-butylbromide — Hyoscine n-butylbromide 10 mg
  Groups: Women with spasmodic syndromes
Drug: Paracetamol — Paracetamol 500 mg
  Groups: Women with spasmodic syndromes

SUMMARY:
What AE occur in routine clinical practice, what is the incidence of AE and Adverse Drug Reaction, how many patients present with AE symptoms related to a potential liver injury. What are the drug utilization patterns in patients, what are the predisposing factors for the occurrence of adverse events and adverse drug reactions.

ELIGIBILITY:
Inclusion criteria:

1. Patients 18 years of age and older who have received at least one dose of BUSCAPINA COMPOSITUM N according to label indications and who attend to one of the pharmacies, clinics, or private doctors office selected for the study.
2. Patients who agree to adhere to the protocol procedures of this study.
3. Women who are not pregnant or breast feeding
4. Persons who sign the informed consent

Exclusion criteria:

1. Patients with allergy to BUSCAPINA COMPOSITUM N or any of the compounds in the formula.
2. Patients with mechanical stenosis of the gastrointestinal tract.
3. Patients with myasthenia gravis.
4. Patients with megacolon.
5. Patients breastfeeding at the time of enrollment or who have become pregnant during treatment with BUSCAPINA COMPOSITUM N.
6. Patients with clinical evidence of immunosuppression.
7. Patients with urinary retention subvesical obstruction (such as prostatic adenoma).
8. Patients with right-angle glaucoma.
9. Patients with tachycardia and tachyarrhythmia.
10. Patients with severe hepatic impairment.
11. Patients with psychiatric disorders.
12. Patients with alcohol dependence or drugs.
13. Patients who discontinue the protocol are not eligible for re-enrollment.
14. Researchers, company personnel or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metropolitan Lima
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Peru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Observational prospective study to evaluate adverse events (AEs), Risk factors and drug utilization of Buscapina Compositum N in adults from metropolitan lima
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended one of 4 specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Buscapina Compositum N: Combination of 10 milligram (mg) of hyoscine n-butylbromide (HBB) and 500 mg of paracetamol. The dose of Buscapina Compositum N was according to label instructions which patients had to acquire on their own (one to two tablets by mouth every 8 hours for 3 to 4 days, swallowed whole with sufficient water).
Period: Overall Study
Arm/Group | Buscapina Compositum N
Started | 360
Completed | 341
Not Completed | 19
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications and who attended to one of the health centers selected for the study.
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications and who attended to one of the health centers selected for the study.
  Years | 36.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications and who attended to one of the health centers selected for the study.
  Participants
    Female | 270
    Male | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Incidence of Adverse Event (AE) Associated to Potential Liver Damage During the Clinical Evaluation of Patients
Description: Percentage of patients with an incidence of Adverse Event (AE) associated to potential liver damage during the clinical evaluation of patients.
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications, attended to one of the health centers selected for the study, and who provided data for the baseline and the follow-up visit.
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 342
Percentage of Patients | 0.0

2. Secondary Outcome: Percentage of Patients With Different Transaminase Levels Found by the Doctor During the Clinical Evaluation of Patients With Symptoms Related to Potential Liver Damage.
Description: Percentage of patients with different transaminase levels found by the doctor during the clinical evaluation of patients with symptoms related to potential liver damage. No patient with symptoms related to potential liver damage was identified, thus analyses of transaminase levels was not performed.
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications, attended to one of the health centers selected for the study, provided data for the baseline and the follow-up visit, and who reported symptoms related to potential liver damage at the follow-up visit.
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 342
Percentage of Patients | NA — No patient with symptoms related to potential liver damage was identified, thus analyses of transaminase levels was not performed.

3. Secondary Outcome: Percentage of Patients With Different Drug Utilization Patterns of Buscapina Compositum N in Patients in Metropolitan Lima
Description: Percentage of patients with different drug utilization patterns of Buscapina Compositum N in patients in Metropolitan Lima.
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 342
Percentage of Patients
  Patient took the medication with liquids (Yes) | 100.0
  Patient took the medication with liquids (No) | 0.0
  Type of liquid used (Water) | 94.7
  Type of liquid used (Juice) | 8
  Type of liquid used (Other) | 2.9
  Amount of liquid used (A straw/sip) | 0.3
  Amount of liquid used (1/4 cup) | 3.8
  Amount of liquid used (1/2 cup) | 33.0
  Amount of liquid used (A full cup) | 44.7
  Amount of liquid used (More than a cup) | 18.1
  Storage of medicine (In a dry and fresh location) | 98.0
  Storage of medicine (In a hot location) | 0.3
  Storage of medicine (In the refrigerator) | 0.0
  Storage of medicine (Other) | 1.8
  Reason - Not taking medicine (No symptoms anymore): number analyzed (Participants) | 107
  Reason - Not taking medicine (No symptoms anymore) | 51.4
  Reason - Not taking medicine (Forgot it): number analyzed (Participants) | 107
  Reason - Not taking medicine (Forgot it) | 23.4
  Reason - Not taking medicine (Had no time): number analyzed (Participants) | 107
  Reason - Not taking medicine (Had no time) | 5.6
  Reason - Not taking medicine (Other): number analyzed (Participants) | 107
  Reason - Not taking medicine (Other) | 12.2
  Reason - Not taking medicine (No answer): number analyzed (Participants) | 107
  Reason - Not taking medicine (No answer) | 7.5

4. Secondary Outcome: Percentage of Patients Per Adverse Event Preferred Term in Patients Who Developed Any Adverse Event During Treatment
Description: Percentage of patients per adverse event preferred term in patients who developed any adverse event during treatment with Buscapina Compositum N.
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications, attended to one of the health centers selected for the study, provided data for the baseline and the follow-up visit, and who developed any adverse event during treatment.
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 342
Percentage of Patients
  Abdominal pain (upper) | 0.3
  Diarrhoea | 0.3
  Nausea | 0.3
  Constipation | 0.3
  Abdominal Pain | 0.3
  Dizziness | 0.3
  Somnolence | 1.2
  Cough | 0.3
  Urine color abnormal | 0.3
  Headache + nausea | 0.3
  Nausea + constipation | 0.3
  Flatulence + constipation | 0.3
  Polydipsia + abdominal pain (upper) | 0.3

5. Secondary Outcome: Percentage of Patients With Different Variables Related to the Occurrence of Increase of Transaminases in Patients Under Treatment With Buscapina Compositum N
Description: Percentage of patients with different variables related to the occurrence of increase of transaminases in patients under treatment with Buscapina Compositum N in Metropolitan Lima. No patient with symptoms related to potential liver damage was identified, thus analyses of transaminase levels was not performed.
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Population: Patients who have received at least one dose of Buscapina Compositum N according to label indications, attended to one of the health centers selected for the study, provided data for the baseline and the follow-up visit.
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscapina Compositum N
Number analyzed (Participants) | 342
Percentage of Patients | NA — No patient with symptoms related to potential liver damage was identified, thus analyses of transaminase levels was not performed

ADVERSE EVENTS:
Time Frame: From the initial dose of study drug until end of the follow up period, up to 113 days
Description: During the observational period, all adverse events following exposure to Buscapina Compositum N were recorded in the case report form, regardless of seriousness or causality.
Arm/Group | Buscapina Compositum N
All-Cause Mortality (participants affected / at risk) | 0/360
Serious Adverse Events (participants affected / at risk) | 0/360
Other Adverse Events (participants affected / at risk) | 0/360

LIMITATIONS AND CAVEATS:
Since the study is conducted at some health centers, it cannot be generalized to the whole population who uses study drug. It is without a control group, thus not able to compare cumulative incidence of AE with the patients not exposed to this drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT02910167/Prot_SAP_000.pdf